CLINICAL TRIAL: NCT07131501
Title: A Single-Arm, Multicenter, Exploratory Clinical Study of Transarterial Chemoembolization (TACE) Combined With Iparomlimab and Tuvonralimab Injection (QL1706) and Lenvatinib for Perioperative Treatment of Resectable Hepatocellular Carcinoma (HCC)
Brief Title: A Single-Arm, Multicenter, Exploratory Clinical Study of TACE Combined With Iparomlimab and Tuvonralimab Injection (QL1706) and Lenvatinib for Perioperative Treatment of Resectable Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xuehao Wang, professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SR-348
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma; Immunotherapy; Preoperative; PD-1; CTLA-4
MeSH Terms: conditions — Carcinoma, Hepatocellular; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Preoperative TACE (1 session) → Iparomlimab and Tuvonralimab Injection (QL1706) + Lenvatinib (Q3W, 2 cycles) → Radical surgery ± intraoperative microwave ablation → Postoperative TACE (1 session) → Iparomlimab and Tuvonralimab Injection (QL1706) (Q3W, ≤17 cycles)
  Interventions: Procedure: Radical surgery; Procedure: TACE treatment; Drug: Iparomlimab and Tuvonralimab Injection (QL1706); Drug: Lenvatinib

INTERVENTIONS:
Procedure: Radical surgery — Radical surgery
Procedure: TACE treatment — TACE treatment (cTACE, Idarubicin): Preoperative: 1 session; Postoperative: 1 session.
Drug: Iparomlimab and Tuvonralimab Injection (QL1706) — Iparomlimab and Tuvonralimab Injection (QL1706): 7.5 mg/kg, intravenous infusion, Day 1 of each cycle, Q3W. Neoadjuvant: 2 cycles; Adjuvant: up to 17 cycles.
Drug: Lenvatinib — Lenvatinib: 8mg (body weight <60kg) or 12mg (body weight ≥60kg), orally (PO), once daily (QD), Q3W. Consistent daily timing. Neoadjuvant: 2 cycles.

SUMMARY:
This is a single-arm, multicenter, exploratory clinical study evaluating the efficacy and safety of TACE combined with Iparomlimab and Tuvonralimab Injection (QL1706) and lenvatinib for perioperative treatment of resectable HCC (CNLC IIb-IIIa excluding Vp3/Vp4 or CNLC Ib-IIa with high-risk recurrence factors). Eligible subjects providing written informed consent will receive study treatment. The primary endpoint is MPR rate.

DETAILED DESCRIPTION:
This is a single-arm, multicenter, exploratory clinical study evaluating the efficacy and safety of TACE combined with Iparomlimab and Tuvonralimab Injection (QL1706) and lenvatinib for perioperative treatment of resectable HCC (CNLC IIb-IIIa excluding Vp3/Vp4 or CNLC Ib-IIa with high-risk recurrence factors). Eligible subjects providing written informed consent will receive study treatment. The primary endpoint is MPR rate.

To standardize TACE efficacy and tolerability, conventional lipiodol-based TACE (cTACE) with idarubicin as the chemotherapeutic agent is employed. The treatment sequence is: Preoperative TACE (1 session) → Iparomlimab and Tuvonralimab Injection (QL1706) + Lenvatinib (Q3W, 2 cycles) → Radical surgery ± intraoperative microwave ablation → Postoperative TACE (1 session) → Iparomlimab and Tuvonralimab Injection (QL1706) (Q3W, ≤17 cycles).

Safety Visits: Occur at screening, pre-TACE, Cycle D1 of neoadjuvant Iparomlimab and Tuvonralimab Injection (QL1706), pre-surgery, pre-postoperative TACE, Cycle D1 of adjuvant Iparomlimab and Tuvonralimab Injection (QL1706), and end of treatment.

Survival Follow-up: Every 12 weeks after safety visits via clinic visit or phone call to collect survival status and subsequent anti-cancer therapy until death, loss to follow-up, sponsor termination, or study completion.

Imaging Assessment: All lesions assessed per RECIST v1.1 and mRECIST. Consistent scanning parameters are required.

Pathological Assessment: Post-surgery assessment of pathological response (MPR, pCR rates) and resection margin status (R0).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate, sign ICF, demonstrate good expected compliance, and be willing to cooperate with follow-up.
2. Age 18-75 years, any gender.
3. HCC diagnosis confirmed by histopathology, cytology, or imaging.
4. Resectable HCC staged as CNLC IIb-IIIa (excluding Vp3 and Vp4) or CNLC Ib-IIa with high-risk recurrence factors, confirmed by multidisciplinary liver surgery expert panel.
5. For CNLC Ib-IIa subjects, presence of at least ONE high-risk recurrence factor.
6. No prior systemic therapy for HCC (chemotherapy, targeted therapy, immunotherapy, etc.). Subjects with prior curative surgery or ablation are eligible only if recurrence occurred >2 years post-resection. Subjects with prior other local therapies are excluded.
7. Child-Pugh class A.
8. ECOG PS score 0-1.
9. Expected survival ≥12 months.
10. Adequate organ function within 7 days prior to study intervention.
11. For subjects with HBV infection.
12. Women of childbearing potential: Must agree to abstinence or use highly effective contraception from ICF signing until ≥120 days after last study drug dose. Negative pregnancy test within 7 days prior to intervention. Not breastfeeding.
13. Male subjects with WOCBP partners: Must agree to abstinence or use highly effective contraception from ICF signing until ≥120 days after last study drug dose. Must not donate sperm during this period. Males with pregnant partners must use condoms.

Exclusion Criteria:

1. Known intrahepatic cholangiocarcinoma, sarcomatoid HCC, mixed carcinoma (>30% ICC component), or fibrolamellar carcinoma. Active malignancy other than HCC within 5 years or concurrently. Cured localized cancers are eligible.
2. Current or history of interstitial lung disease/pneumonitis requiring steroids, or other active lung disease potentially interfering with immune-related pulmonary toxicity evaluation/management, or active pneumonia/severe impaired pulmonary function on screening CT. Active tuberculosis.
3. Active autoimmune disease or history of autoimmune disease with potential recurrence. Vitiligo, psoriasis, alopecia not requiring systemic therapy, controlled Type I diabetes on insulin, or childhood asthma resolved in adulthood without intervention are eligible. Asthma requiring bronchodilators is excluded.
4. Systemic immunosuppressive therapy (>10 mg/day prednisone equivalent) within 2 weeks prior to intervention.
5. Active infection, unexplained fever ≥38.5°C within 1 week prior, or baseline WBC >15 × 10⁹/L. Therapeutic antibiotics (IV/oral) within 2 weeks prior (prophylactic IV antibiotics ≤48h duration allowed).
6. Primary or acquired immunodeficiency.
7. Live attenuated vaccine within 4 weeks prior to intervention or anticipated need during study or within 60 days after last Iparomlimab and Tuvonralimab Injection dose.
8. Significant bleeding symptoms or predisposition within 6 months prior. If baseline fecal occult blood positive, repeat test; if still positive, requires gastroscopy.
9. Known hereditary/acquired bleeding/thrombotic diathesis. Current therapeutic-dose anticoagulants/thrombolytics (prophylactic low-dose aspirin allowed).
10. Arterial thromboembolic events within 6 months prior.
11. Poorly controlled cardiac disease.
12. Hypertension uncontrolled by medication (average SBP ≥140 mmHg or DBP ≥90 mmHg on ≥2 readings). History of hypertensive crisis or encephalopathy.
13. Major vascular disease within 6 months prior.
14. Serious unhealed wounds, active ulcers, or untreated fractures.
15. Major surgery within 4 weeks prior or anticipated major surgery during study.
16. Inability to swallow pills, malabsorption syndrome, or GI condition affecting absorption.
17. Bowel obstruction or related symptoms/signs within 6 months prior requiring parenteral support/feeding. Subjects with prior resolved obstruction treated definitively (surgically) may be eligible after assessment.
18. Strong CYP3A4 inducers within 2 weeks prior or strong CYP3A4 inhibitors within 1 week prior.
19. Known hypersensitivity to any study drug or excipient.
20. Participation in another investigational drug study within 4 weeks prior.
21. Pregnancy or lactation.
22. Any other condition deemed unsuitable by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-08-11 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) rate | 60-day
  Proportion of subjects achieving MPR (defined as ≤10% residual viable tumor cells in the original tumor bed after neoadjuvant therapy, i.e., ≥90% necrosis) among all enrolled subjects.

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) rate | 60-day
  Proportion of subjects achieving pCR (defined as no residual viable tumor cells in the original tumor bed after neoadjuvant therapy) among all enrolled subjects.
R0 resection rate | 60-day
  R0 resection rate
Objective Response Rate (ORR) | 6-month
  Proportion of subjects achieving Complete Response (CR) or Partial Response (PR) among all enrolled subjects (assessed by investigators per RECIST v1.1 and mRECIST).
Disease Control Rate (DCR) | 6-month
  Proportion of subjects achieving CR, PR, or Stable Disease (SD) among all enrolled subjects (assessed by investigators per RECIST v1.1 and mRECIST)
Event-Free Survival (EFS) | 3-year
  Time from the start of neoadjuvant therapy to the first occurrence of any of the following events: disease progression precluding surgery, postoperative recurrence or metastasis, or death from any cause.
Recurrence-Free Survival (RFS) | 3-year
  (For patients undergoing Radical surgery only) Time from the date of Radical surgery to tumor recurrence or death from any cause, whichever occurs first.
Overall Survival (OS) | 3-year
  Time from the start of neoadjuvant therapy to death from any cause.
Adverse event (AE) | 3-year
  Adverse events (AEs), Serious Adverse events (SAEs), surgery related safety.

CONTACTS AND LOCATIONS:
Overall Officials: Xuehao Wang, Study Chair — The First Affiliated Hospital with Nanjing Medical University; Yongxiang Xia, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No